CLINICAL TRIAL: NCT07182942
Title: The Effect and Mechanism of Xiqing Regulating Intestinal Homeostasis on Drug Efficacy of Chronic Kidney Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chujin Cao (Other)
Responsible Party: Sponsor-Investigator, Chujin Cao, associated professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 103630
Record Dates: First submitted 2025-09-08; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: CKD; Drug Effect
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CKD+Xiqing (Experimental): This group is experimental one, which is CKD patients with Xiqing intervention alone.
  Interventions: Drug: Xiqing
- CKD+Pro (Experimental): This group is experimental one, which is CKD patients with the probiotics intervention alone.
  Interventions: Drug: probiotics
- CKD+Xiqing+Pro (Experimental): This group is experimental one, which is CKD patients with the intervention of Xiqing combined the probiotics.
  Interventions: Drug: Xiqing; Drug: probiotics

INTERVENTIONS:
Drug: Xiqing — oral intervention of Xiqing
  Arms: CKD+Xiqing; CKD+Xiqing+Pro
Drug: probiotics — oral intervention of probiotics
  Arms: CKD+Pro; CKD+Xiqing+Pro

SUMMARY:
Chronic kidney disease (CKD) has become a major public health problem worldwide. Patients with CKD are often accompanied by azotemia due to impaired renal function and excretion of nitrogen metabolic waste, which leads to multiple organ dysfunction, cardiac dysfunction and other complications. Therefore, it is an important strategy in the treatment of CKD to reduce the burden of kidney in CKD patients by removing nitrogen metabolic wastes in the body. Xiqing, which includes coated aldehyde oxystarch capsules, is a drug with adsorption effect. As an effective nitrogen metabolic waste adsorbent, it is widely used in the treatment of CKD patients. Gut is an important organ for the generation of nitrogen metabolic waste in the body. Intestinal homeostasis is an important regulator of nitrogen metabolism, and supplementation of probiotics is one of the main ways to regulate intestinal homeostasis. A study published by the team of investigators in the journal Cell Metabolism in 2021 confirmed that probiotics (Lactobacillus casei Zhang) reduced the BUN level in CKD mice, intestinal inflammation and the permeability of intestinal mucosal barrier, and delay the progression of CKD patients through animal experiments and clinical trials. So, whether the application of Xiqing changes intestinal homeostasis, including intestinal flora structure, function and function of intestinal mucosa, intestinal metabolites? Whether drug effect is affected by intestinal balance of CKD? What is the mechanism? Is Xiqing combined with probiotics more conducive to reducing BUN level and delaying the progression of CKD patients? The discussion of the problem and solution will help clinicians for the pioneering understanding of the use of Xiqing.

In this study, the investigators designed a prospective, randomized, open-label, blinded end-point clinical trial, using microbial diversity, metagenomics, targeted and non-targeted metabolomics detection and other technologies, through the joint analysis of multi-omics data, to explore the effect of the use of Xiqing on the intestinal homeostasis of CKD, and the extent of the drug efficacy of Xiqing is affected by the intestinal homeostasis of CKD. The effect of Xiqing combined the probiotics regulating intestinal homeostasis on CKD and the molecular mechanism, which provide more research references for the clinical application of Xiqing.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent was obtained;
2. ranging in age from 18 to 75 years;
3. CKD stage 3-5, that is, eGFR < 60 mL/min/1.73 m2 with non-dialysis stage, no dialysis indication, temporarily stable condition and drug control stage;
4. tolerance of Xiqing and probiotics treatment.

Exclusion Criteria:

1. with severe active infection, influence of nutritional status in patients with malignant tumor and other diseases;
2. patients during pregnancy or lactation;
3. unstable vital signs, the condition is not stable, need dialysis patients;
4. patients with intolerance of Xiqing;
5. patients with intolerance of probiotics;
6. taking corticosteroids, antibiotics or other immunosuppressive agents within the past 3 months;
7. taking adsorbent drugs, such as medicinal charcoal tablets, within the past 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Kidney disease progression | 3 months
  Entry into end-stage renal disease or serum creatinine values doubled

SECONDARY OUTCOMES:
Cardiovascular events | 3 months
  Occurrence of cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yao, PhD, Study Director — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China